CLINICAL TRIAL: NCT03165253
Title: The Effects of the Synbiotic "Bifidobacterium Lactis B94 Plus Inulin" Addition on Standard Triple Therapy of Helicobacter Pylori Eradication in Children
Brief Title: The Effects of a Synbiotic Addition on Eradication Therapy of Helicobacter Pylori Infection in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gonca Handan Ustundag, Associate Professor of Pediatrics, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-10-08/03
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori infection; Children; Synbiotic; Standard Triple Therapy
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic Group (Active Comparator): The patients will be treated with the standard triple therapy that consists of amoxicillin oral tablet 50 mg/kg/d and clarithromycin oral tablet 15 mg/kg/d twice daily for 14 days, and omeprazole 1 mg/kg/d once daily for a month, and the synbiotic Bifidobacterium animalis oral product (5000000000 colony forming units/dose) plus inulin (900 mg) given a single dose for 14 days, concurrently.
  Interventions: Drug: Bifidobacterium Animalis Oral Product; Drug: Amoxicillin Oral Tablet; Drug: Clarithromycin Oral Tablet; Drug: Omeprazole
- Standard Therapy Group (Other): The patients in this group will be treated with standard triple therapy only. The standard triple therapy consists of amoxicillin oral tablet 50 mg/kg/d and clarithromycin oral tablet 15 mg/kg/d twice daily for 14 days, and omeprazole 1 mg/kg/d once daily for a month.
  Interventions: Drug: Amoxicillin Oral Tablet; Drug: Clarithromycin Oral Tablet; Drug: Omeprazole

INTERVENTIONS:
Drug: Bifidobacterium Animalis Oral Product — The synbiotic group will receive this product.
  Other Names: Bifidobacterium lactis
  Arms: Synbiotic Group
Drug: Amoxicillin Oral Tablet — 50mg/kg/day B.I.D.
  Other Names: Amoxicillin
Drug: Clarithromycin Oral Tablet — 15 mg/kg/day B.I.D.
  Other Names: Clarithromycin
Drug: Omeprazole — 1 mg/kg/day
  Other Names: Omeprazole Capsule

SUMMARY:
The aim of the study is to evaluate the effects of the synbiotic Bifidobacterium animalis ssp. lactis B94 plus inulin addition to the standard triple therapy on Helicobacter pylori infection eradication rates in children.

DETAILED DESCRIPTION:
The study aims to evaluate the effects of the synbiotic Bifidobacterium animalis ssp. lactis B94 plus inulin addition to the standard triple therapy on the eradication rates of Helicobacter pylori (H. pylori) infection in children. The subjects are children between 6 to 16 years old who had biopsy proven H. pylori infection. The subjects will be randomly classified into two groups. The first group will receive the standard triple therapy consisting of amoxicillin oral tablet (50 mg/kg/day) + clarithromycin oral tablet (15 mg/kg/day) + omeprazole oral capsule (1mg/kg/day). The second group will receive the standard triple therapy and Bifidobacterium animalis ssp. lactis B94 (5000000000 colony forming units/dose) plus inulin (900 mg) containing sachet for 14 days, concurrently. Eradication will be determined by 14-Carbon-urea breath test 4-6 weeks after therapy discontinuation. The eradication rates, the occurrence of side effects and the alterations of initial symptoms will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Children who are investigated by a standard esophagogastroduodenoscopy (EGD) for gastrointestinal symptoms those suggesting of an organic disease such as chronic abdominal pain, unexplained nausea and/or vomiting, severe regurgitation, gastrointestinal bleeding, unexplained weight loss, or chronic diarrhea and who are found to be H. pylori positive in gastric biopsies are included in the study.

Exclusion Criteria:

* Patients who were treated for H. pylori infection previously, or who used an antimicrobial agent, bismuth, a non-steroid anti-inflammatory drug, or any form of gastric acid suppressor during the eight weeks prior to EGD, or who had history of major gastrointestinal surgery, chronic renal or hepatic disease and who were known to have drug allergy were excluded from the study.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The eradication rates | 4-6 weeks after cessation of treatment
  The eradication of H. pylori infection will be assessed by 14-carbon-urea breath test and the difference between eradication rates will be compared between the study groups.

SECONDARY OUTCOMES:
The eradication therapy associated side effects | 14 days period during the treatment
  Patients will be monitored at clinical visits and will be asked to recall for any side effects during the treatment protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca H Ustundag, MD, Principal Investigator — Associate professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Koletzko S, Jones NL, Goodman KJ, Gold B, Rowland M, Cadranel S, Chong S, Colletti RB, Casswall T, Elitsur Y, Guarner J, Kalach N, Madrazo A, Megraud F, Oderda G; H pylori Working Groups of ESPGHAN and NASPGHAN. Evidence-based guidelines from ESPGHAN and NASPGHAN for Helicobacter pylori infection in children. J Pediatr Gastroenterol Nutr. 2011 Aug;53(2):230-43. doi: 10.1097/MPG.0b013e3182227e90. PMID 21558964
- [Result] Gotteland M, Brunser O, Cruchet S. Systematic review: are probiotics useful in controlling gastric colonization by Helicobacter pylori? Aliment Pharmacol Ther. 2006 Apr 15;23(8):1077-86. doi: 10.1111/j.1365-2036.2006.02868.x. PMID 16611267
- [Derived] Ustundag GH, Altuntas H, Soysal YD, Kokturk F. The Effects of Synbiotic "Bifidobacterium lactis B94 plus Inulin" Addition on Standard Triple Therapy of Helicobacter pylori Eradication in Children. Can J Gastroenterol Hepatol. 2017;2017:8130596. doi: 10.1155/2017/8130596. Epub 2017 Jun 1. PMID 28656129